CLINICAL TRIAL: NCT06757634
Title: VIKTORIA-2: A Randomized, Open-Label, Phase 3 Study of Fulvestrant and CDK4/6 Inhibitors With or Without Gedatolisib as First-Line Treatment in Patients With HR-Positive and HER2-Negative Advanced Breast Cancer
Brief Title: Phase 3 Study of Gedatolisib as First-Line Treatment for Patients With HR-Positive, HER2-Negative Advanced Breast Cancer (VIKTORIA-2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celcuity Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELC-G-302
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer, Advanced or Metastatic; Gedatolisib; HR Positive; ER Positive; HER2 Negative; PIK3CA MT; PI3K
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — palbociclib; ribociclib; Fulvestrant; gedatolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Gedatolisib + Palbociclib or Ribociclib + Fulvestrant (Experimental): Drug: Gedatolisib Participants will receive intravenous (IV) gedatolisib once weekly for 3 weeks (Days 1, 8, 15) followed by 1 week off
  Interventions: Drug: Arm A: Gedatolisib + Palbociclib or Ribociclib + Fulvestrant; Drug: Arm B: Palbociclib or Ribociclib + Fulvestrant
- Arm B: Palbociclib or Ribociclib + Fulvestrant (Active Comparator): Drug: Palbociclib Participants will receive oral palbociclib on Days 1-21 of each 28-day cycle
  Interventions: Drug: Arm A: Gedatolisib + Palbociclib or Ribociclib + Fulvestrant; Drug: Arm B: Palbociclib or Ribociclib + Fulvestrant

INTERVENTIONS:
Drug: Arm A: Gedatolisib + Palbociclib or Ribociclib + Fulvestrant — Drug: Gedatolisib Participants will receive intravenous (IV) gedatolisib once weekly for 3 weeks (Days 1, 8, 15) followed by 1 week off
  Other Names:
  • PF-05212384 Drug: Palbociclib Participants will receive oral palbociclib on days 1-21 of each 28-day cycle.
  Other Names:
  • IBRANCE Drug: Ribociclib Participants will receive oral ribociclib on Days 1-21 of each 28-day cycle
  Other Names:
  • KISQALI® Drug: Fulvestrant Participants will receive intramuscular (IM) fulvestrant every 2 weeks during Cycle 1 and then every 4 weeks
  Other Names:
  • Faslodex
  Other Names: PF-05212384, IBRANCE, KISQALI®, Faslodex
Drug: Arm B: Palbociclib or Ribociclib + Fulvestrant — Drug: Palbociclib Participants will receive oral palbociclib on Days 1-21 of each 28-day cycle
  Other Names:
  • IBRANCE Drug: Ribociclib Participants will receive oral ribociclib on Days 1-21 of each 28-day cycle
  Other Names:
  • KISQALI®
  Drug: Fulvestrant Participants will receive intramuscular (IM) fulvestrant approximately every 2 weeks during Cycle 1 then approximately every 4
  Other Names:
  • Faslodex
  Other Names: IBRANCE, KISQALI®, Faslodex

SUMMARY:
This is a Phase 3, open-label, randomized, clinical trial evaluating the efficacy and safety of gedatolisib plus fulvestrant and CDK4/6 Inhibitors for the treatment of patients with locally advanced or metastatic HR+/HER2- advanced breast cancer.

DETAILED DESCRIPTION:
This is a Phase 3, open-label, randomized clinical trial evaluating the efficacy and safety of gedatolisib plus fulvestrant combined with a CDK4/6 inhibitor (Investigator's choice of palbociclib or ribociclib) for the treatment of patients with advanced (inoperable) or metastatic hormone receptor positive, human epidermal growth factor receptor 2 negative (HR+/HER2-) breast cancer whose disease has progressed during or within 12 months of adjuvant treatment with endocrine therapy (either an AI or tamoxifen), and who have not received prior systemic therapy for ABC. Gedatolisib is an intravenously administered pan-PI3K/mTOR inhibitor. Palbociclib is a CDK4/6 inhibitor. Fulvestrant is a selective estrogen receptor degrader (SERD). Following completion of the safety run-in phase to determine the gedatolisib dose with ribociclib, subjects will be assigned to 1 of 2 cohorts based on their PIK3CA status and then randomized to either the investigational treatment arm (gedatolisib with fulvestrant and ribociclib or palbociclib) or standard-of-care control arm (fulvestrant and ribociclib or palbociclib).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of metastatic or locally advanced HR+/HER2- breast cancer
2. Adult females, pre- and/or post-menopausal, and adult males. Pre-menopausal (and peri-menopausal) women can be enrolled if amenable to treatment with an LHRH agonist. Patients are to have commenced concomitant treatment with LHRH agonist prior to or on Cycle 1, Day 1 and must be willing to continue for the duration of the study.
3. Negative pregnancy test for females of childbearing potential. Female subjects who are not surgically sterile must use a medically effective contraceptive method from screening until 2 years after the last dose of study treatment.
4. Progression of disease during or within 12 months of completing (neo)adjuvant ET.
5. Adequate archival, fresh tumor tissue, or liquid biopsy for the analysis of PIK3CA mutational status.
6. Permitted prior therapies:

   1. (neo)adjuvant fulvestrant or any selective ER degrader only if the treatment duration < 6 months
   2. (neo)adjuvant chemotherapy
   3. (neo)adjuvant CDK4/6 inhibitor, unless PD was on or within 6 months of discontinuation of CDK4/6i
7. Subject has radiologically measurable disease according to RECIST v1.1, per local assessment. Patients with evaluable bone-only disease are not eligible. Patients with bone-only disease that has lytic or mixed lytic/blastic lesions and at least one measurable soft tissue component per RECIST v1.1 may be eligible.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
9. Life expectancy of at least >6 months.
10. Adequate bone marrow, hepatic, renal and coagulation function.

Exclusion Criteria:

1. Concurrent malignancies other than adequately treated non-melanoma skin cancer. Previous malignancies in remission but curatively treated with no evidence of disease progression and judged by local Investigator to be at low risk of impacting health or survival while on study.
2. Prior treatment with a phosphoinositide 3-kinase (PI3K) inhibitor, a protein kinase B (Akt) inhibitor, or a mechanistic target of rapamycin (mTOR) inhibitor
3. Prior treatment with systemic anticancer therapy for ABC
4. Subjects with type 1 diabetes
5. Known and untreated, or active, brain or leptomeningeal metastases
6. History of clinically significant cardiovascular abnormalities
7. History of drug-induced symptomatic interstitial lung disease (pneumonitis) or hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization to the date of death due to any cause, up to approximately 48 months
  Progression Free Survival (PFS) in Patients with PIK3CA ND and PIK3CA MT Breast Cancer
  PFS is defined as the time from randomization to death or the first documented progression, whichever occurs first, confirmed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria, as determined based on blinded independent central review (BICR)

SECONDARY OUTCOMES:
Overall Survival (OS) in Patients with PIK3CA ND and PIK3CA MT Breast Cancer | From date of randomization to the date of death due to any cause, up to approximately 48 months
  OS is defined as the length of time from randomization until the date of death from any cause method, where PFS is defined as the time from randomization to death or the first documented progression, whichever occurs first, confirmed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria, as determined based on blinded independent central review (BICR)
Overall Response Rate (ORR) in Patients with PIK3CA ND and PIK3CA MT Breast Cancer | Up to approximately 48 months
  Percentage of subjects who achieved an objective response according to RECIST v1.1 criteria (complete response [CR] or partial response [PR]) as assessed by BICR)
Overall Response Rate (ORR) in Patients with PIK3CA ND and PIK3CA MT Breast Cancer | Up to approximately 48 months
  Percentage of subjects who achieved an objective response according to RECIST v1.1 (CR or PR) as assessed by BICR
Duration of Response (DOR) in Patients with PIK3CA ND and PIK3CA MT Breast Cancer | Up to approximately 48 months
  Time from the assessment of initial response (PR or better) to death or first documented radiologically confirmed disease progression as assessed by BICR, whichever occurs first
Time to Response (TTR) in Patients with PIK3CA ND and PIK3CA MT Breast Cancer | Time from randomization to the first assessment of PR or better as assessed by BICR
  Time to Response (TTR) in Patients with PIK3CA ND and PIK3CA MT Breast Cancer
Clinical Benefit Rate (CBR) in Patients with PIK3CA ND and PIK3CA MT Breast Cancer | Up to approximately 48 months
  Percentage of subjects with CR or PR; or with stable disease (SD) lasting >24 weeks as assessed by BICR
Quality of Life (QOL) Functional Assessment of Cancer Therapy - Breast Trial Outcome Index (FACT-B TOI) | From baseline to 30 Day Safety Follow-up
  Questions in Patients with PIK3CA ND and PIK3CA MT Breast Cancer
Adverse Events | Up to approximately 48 months
  Type, incidence, severity (as graded by the NCI CTCAE v5.0), seriousness, and relationship to study medications of Adverse Events and any laboratory abnormalities in Arm A compared with Arm B

CONTACTS AND LOCATIONS:
Locations (203):
- United States (22):
  - City of Hope Medical Center, Duarte, California
  - Providence Medical Foundation, Fullerton, California
  - UCLA Hematology Oncology Santa Monica, Los Angeles, California
  - BRCR Medical Center, Inc- Internal Medicine, Plantation, Florida
  - BRCR Medical Center, INC, Tamarac, Florida
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Mercy Health-Paducah Cancer Center, Paducah, Kentucky
  - American Oncology Partners, P.A., Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Washington University School of Medicine in Saint Louis, St Louis, Missouri
  - SCL Health - Cancer Centers of Montana, Billings, Montana
  - Weill Cornell Medical College - NewYork-Presbyterian Hospital, New York, New York
  - Clinical Research Alliance, Inc., Westbury, New York
  - Stefanie Spielman Comprehensive Breast Center at Olentangy River Road, Columbus, Ohio
  - Rittenhouse Hematology/Oncology, Philadelphia, Pennsylvania
  - Sanford Health, Sioux Falls, South Dakota
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Mays Cancer Center, San Antonio, Texas
  - Bon Secours St. Francis Medical Oncology Center, Midlothian, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Argentina (13):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA, Buenos Aires
  - Pergamino Clinic, Buenos Aires
  - CENIT Foundation, Buenos Aires
  - Fleischer Medical Center (Centro Medico Fleischer), Buenos Aires
  - Fundacion Respirar, Buenos Aires
  - Centro Oncológico Korben, Buenos Aires
  - Alexander Fleming Institute, Buenos Aires
  - Center for Medical Education and Clinical Research (CEMIC), Buenos Aires
  - Cordoba Oncology Institute (IONC), Córdoba
  - Centro Oncologico de Excelencia, La Plata
  - Fundación CORI, La Rioja
  - Center of Nuclear and Molecular Medicine of Entre Rios (CEMENER), Paraná
  - Rosario's Oncology Institute and Medical Specialities (IOR), Rosario
- Australia (6):
  - GenesisCare - St Andrews, Adelaide
  - Breast Cancer Research Centre, Nedlands
  - Icon Cancer Centre Southport, Southport
  - Sydney Adventist Hospital, Wahroonga
  - Westmead Hospital, Westmead
  - The Queen Elizabeth Hospital, Woodville
- Belgium (5):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hopital De Charleroi, Charleroi
  - Universitair Ziekenhuis Gent - Medische Oncologie, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse - Medische Oncologie, Hasselt
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Brazil (11):
  - CTO Centro de Tratamento Oncológico, Belém
  - Oncocentro Belo Horizonte, Belo Horizonte
  - Centro Regional Integrado de Oncologia - CRIO, Fortaleza
  - Pronutrir Oncologia e Nutrição, Fortaleza
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia LTDA, Ijuí
  - Catarina Pesquisa Clinica, Itajaí
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto
  - Bahia Oncology Center, Salvador
  - Hospital A.C.Camargo, São Paulo
  - Instituto D'or de Pesquisa e Ensino - ONCO STAR, São Paulo
- Bulgaria (6):
  - Complex Oncology Center - Burgas, Burgas
  - Multi-profile Hospital For Active Treatment-Uni Hospital Ltd., Panagyurishte
  - Complex Oncological Centre Ruse, Rousse
  - MHAT Nadezhda - Medical Oncology Clinic, Sofia
  - MHAT "Serdika" EOOD, Base 2 - Second Department of Medical Oncology, Sofia
  - USHAT of Oncology, Sofia
- Czechia (7):
  - Masarykuv onkologicky ustav - Oddeleni klinickych hodnoceni, Brno
  - Multiscan s.r.o. - Ambulance klinicke onkologie se stacionarem, Hořovice
  - FN Hradec Kralove - Klinika onkologie a radioterap, Hradec Králové
  - Fakultni nemocnice Olomouc - Onkologicka klinika, Olomouc
  - FN Kralovske Vinohrady - Radioterapeuticka a onkologicka klinika, Prague
  - Fakultni Thomayerova Nemocnice - Onkologicka klinika, Prague
  - Fakultni Nemocnice v Motole, Prague
- France (9):
  - Centre Hospitalier Universitaire D'Amiens (Hopital Sud) - Oncologie Medicale - Cancerolo, Amiens
  - Centre Georges François Baclesse, Caen
  - Centre Georges Francois Leclerc - service d'oncologie médicale, Dijon
  - Clinique Victor Hugo / Centre Jean Bernard, Le Mans
  - CHU La Timone, Marseille
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers - Médico-Chirurgical De Cardiol, Poitiers
  - Centre de Lutte Contre le Cancer (CLCC) - Institut de Cancerologie de l'Ouest (ICO) - Rene Gauducheau - Oncology, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Universitätsklinikum Düsseldorf - Gynecology, Düsseldorf
  - Universitätsmedizin Johannes Gutenberg, Mainz
  - CaritasKlinikum Saarbrücken St. Theresia, Saarbrücken
  - Helios Klinikum Wuppertal, Wuppertal
- Greece (7):
  - Areteio Hospital, Athens
  - University General Hospital of Heraklion, Heraklion
  - Iaso Thessalia General Clinic Private Obstetrics S.A., Larissa
  - General University Hospital Of Larissa, Larissa
  - Metropolitan Hospital, Piraeus
  - Athens Medical Center S.A., Thessaloniki
  - Theageneio Cancer Hospital, Thessaloniki
- Hungary (6):
  - Debreceni Egyetem Klinikai Központ Nagyerdei Campus - Onkológiai Klinika, Debrecen
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktatokorhaz, Győr
  - Békés Megyei Központi Kórház Pándy Kálmán Tagkórház - Oncology, Gyula
  - Bacs-Kiskun Varmegyei Oktatakorhaz, Kecskemét
  - University of Pecs- Oncology Dept., Pécs
  - Tolna Varmegyei Balassa Janos Korhaz, Szekszárd
- Italy (15):
  - Presidio Ospedaliero S. Croce - Oncologia, Fano
  - IRCCS Ospedale Policlinico San Martino - Clinica di Oncologia Medica, Genova
  - IRST IRCCS - Oncologia Medica, Meldola
  - IEO - Istituto Europeo di Oncologia, IRCCS, Milan
  - Istituto Clinico Humanitas, Milan
  - AOU di Modena, Policlinico di Modena - Attività Integrata di Oncologia ed Ematologia, Modena
  - Istituto Nazionale dei Tumori - Fondazione Pascale, IRCCS, Napoli
  - Ospedale Maggiore, AOU Parma, Parma
  - IRCCS Policlinico San Matteo, Università degli studi di Pavia, Pavia
  - Ospedale "Santa Maria delle Croci" di Ravenna - Oncologia, Ravenna
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
  - Umberto I Policlinico di Roma, Università La Sapienza, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - Borgo Trento, Ospedale Civile Maggiore, AOU Integrata Verona, Verona
- Malaysia (7):
  - Penang Adventist Hospital, George Town
  - Hospital Universiti Sains Malaysia, Kota Bharu
  - Hospital Kuala Lumpur - Surgery, Kuala Lumpur
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - Beacon Hospital, Petaling Jaya
  - National Cancer Institute - Radiotherapy and Oncology, Putrajaya
- Mexico (7):
  - San Peregrino Unidad de Investigacion, Aguascalientes
  - Office of Emanuel de la Mora Jimenez, MD/equiv, Guadalajara
  - Clinical Research Center Chapultepec Mexico City, Mexico City
  - Centro de Atencion Oncologica Viva, Mexico City
  - Avix Clinical Research, Monterrey
  - Filios High Medicine, Monterrey
  - Administrative Society of Health Services, SC, Morelia
- Poland (8):
  - Centrum Onkologii im. prof. F. Lukaszczyka - Ambulatorium Chemioterapii, Bydgoszcz
  - Przychodnia Lekarska KOMED, Konin
  - Pratia MCM Kraków, Krakow
  - Instytut Medyczny Santa Familia, Lodz
  - SP ZOZ Opolskie Centrum Onkologii - Oddzial Onkologii Klinicznej z Odcinkiem Dziennym, Opole
  - Zachodniopomorskie Centrum Onkologii - Osrodek Innowacyjnosci, Rozwoju i Badan Klinicznych, Szczecin
  - LUX MED Onkologia Sp. z o.o., Szpital Szamocka - Oddzial Onkologii Klinicznej/Chemioterapii, Warsaw
  - Narodowy Instytut Onkologii im. Marii SkÅ'odowskiej-Curie â€" PaÅ"stwowy Instytut Badawczy - Klinika Nowotworow Piersi i Chirurg, Warsaw
- Portugal (6):
  - Centro Hospitalar e Universitário de Coimbra, Coimbra
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil - Oncologia Medica, Lisbon
  - Hospital da Luz de Lisboa - Learning Health, Lisbon
  - H. de Santa Maria. Centro Hospitalar Lisboa Norte - Oncologia, Lisbon
  - Hospital CUF Descobertas, Lisbon
  - Centro Hospitalar Universitario do Porto - H. Santo Antonio, Porto
- Romania (8):
  - Centrul de Oncologie Sf Nectarie - Medical Oncology, Baia Mare
  - Oncopremium Team - Medical Oncology, Baia Mare
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Bucharest
  - Institutul Oncologic Prof Dr Alexandru Trestioreanu Bucuresti, Cluj-Napoca
  - Onco Clinic Consult, Craiova
  - Radiotherapy Center Cluj, Floreşti
  - Centrul de Oncologie Euroclinic, Iași
  - Institutul Regional de Oncologie Iasi - Medical Oncology, Iași
- South Korea (13):
  - National Cancer Center - Breast Cancer, Goyang
  - Gachon University Gil Medical Center - Oncology, Incheon
  - CHA Bundang Medical Center - Oncology, Seongnam-si
  - Korea University Anam Hospital - Gastroenterological Surgery, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System, Severance hospital, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center - Hematology & Oncology, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital - Hematology and Oncology, Seoul
  - Ajou University Hospital - Hematology/Oncology, Suwon
  - Ulsan University Hospital, Ulsan
- Spain (13):
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Del Mar, Barcelona
  - Hospital Clinic De Barcelona, Barcelona
  - Caceres Hospital Complex - San Pedro de Alcantara General Hospital, Cáceres
  - Hospital Clínico Universitario Virgen De La Arrixaca, El Palmar
  - Institut Catala D'oncologia, L'Hospitalet de Llobregat
  - H.U Arnau De Vilanova Lleida, Lleida
  - Hospital Beata Maria Ana de Jesus, Madrid
  - Hospital Universitario Ramon y Cajal - Oncología Médica, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Complejo Hospitalario Universitario De Santiago, Santiago de Compostela
  - Fundacion Instituto Valenciano de Oncologia, Valencia
- Taiwan (11):
  - Changhua Christian Medical Foundation - Changhua Christian Hospital - Neurology, Changhua
  - National Taiwan University Hospital - Yunlin Branch - Oncology, Douliu
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital - Breast Surgery, Kaohsiung City
  - China Medical University Hospital - Breast Surgery, Taichung
  - Taichung Veterans General Hospital - General Surgery, Taichung
  - National Cheng Kung University Hospital - Gynecology/Obstetrics, Tainan
  - Chi Mei Medical Center - YongKang - Oncology and Hematology, Tainan
  - National Taiwan University Hospital - Oncology, Taipei
  - Taipei Medical University - Shuang Ho Hospital Ministry of Health and Welfare - Nephrology, Taipei
  - Taipei Veterans General Hospital - Hematology, Taipei
  - Taipei Municipal Wanfang Hospital - Managed by Taipei Medical University - Hematology and Oncology, Taipei
- Thailand (5):
  - King Chulalongkorn Memorial Hospital [Medical Oncology], Bangkok
  - Rajavithi Hospital, Bangkok
  - Siriraj Hospital - Medical Oncology, Bangkok
  - Prince of Songkla University - Internal Medicine, Hat Yai
  - Banphaeo General Hospital, Samut Sakhon
- Turkey (Türkiye) (14):
  - Adana Baskent Practice and Research Hospital - Oncology, Adana
  - Gulhane Training and Research Hospital - Medical Oncology, Ankara
  - Hacettepe University Medical Faculty - Hematology, Ankara
  - Dr Abdurrahman Yurtaslan Training and Research Hospital - Medical Oncology, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Ankara University Medical Faculty - Oncology, Ankara
  - Dicle University Medical Faculty Hospital Medical Oncology, Diyarbakır
  - Trakya University Medical Faculty - Oncology, Edirne
  - Medical Park Hastaneler Grubu - I.A.U. VM Medical Park Florya, Istanbul
  - Medipol Mega Hospital - Medical Oncology, Istanbul
  - Istanbul Goztepe Prof. Dr. Suleyman Yalcin City Hospital - Medical Oncology, Istanbul
  - Kocaeli Uni Egt ve Uyg Hast, İzmit
  - Necmettin Erbakan University Meram Medical Faculty - Oncology, Konya
  - VM Medical Park Mersin Hastanesi, Mezitli

IPD SHARING:
Plan to Share IPD: Undecided